CLINICAL TRIAL: NCT03176602
Title: Combining Two Commonly Adopted Nutrition Instruments in the Critical Care Setting is Superior to Administering Either One Alone
Brief Title: Prognostic Value of the SGA and NUTRIC in the ICU
Status: Completed | Type: Observational
Sponsor: JurongHealth (Other Government)
Collaborators: Flinders University (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/00878/1
Record Dates: First submitted 2017-06-02; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Critical Illness; Malnutrition
Keywords: Subjective Global Assessment; Nutrition Risk in Critically ill Score; Critical Illness
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients admitted to the ICU: All patients ≥ 18 years old who had ≥ 24 hours length of stay in the ICU

SUMMARY:
There are two nutrition assessment tools that are commonly used in the ICU, namely the Subjective Global Assessment (SGA) and Modified Nutrition Risk in Critically Ill Score (mNUTRIC). It has been proposed that both assessments should be performed in the ICU but their combined prognostic ability has not been adequately assessed.

This study aimed to: 1) determine the agreement between SGA and mNUTRIC scores, and 2) quantify their utility in discriminating and quantifying hospital mortality risk both independently and in combination.

DETAILED DESCRIPTION:
This prospective observational study will be conducted in a 35-bed mixed ICU in Ng Teng Fong General Hospital, and all the intensivists and nurses will be blinded to the objectives of the study. All patients admitted to the ICU will be consecutively included in the study. For patients readmitted to the ICU during the same hospitalisation, only data from the first admission will be collected.

As per routine care, all patients will have their nutritional status assessed by the dietitian within 48 hours of ICU admission. Information required for the nutritional assessment (SGA) will be obtained from the patients or their main care givers, and nutritional status will be dichotomized into well-nourished and malnourished.

The electronic medical records automatically and prospectively collects all data required to calculate the mNUTRIC. At the end of the study, the mNUTRIC will be retrospectively calculated. Patients with values of "0-4" will be classified as low-mNUTRIC and "5-9" as high-mNUTRIC.

The primary outcome will be hospital mortality and all patients will be followed until discharge or death, for up to one year after admission to the ICU.

Agreement and mortality discriminative value (i.e. discrimination) of the 2-category classification of mNUTRIC (Low- and high-mNUTRIC) and SGA (SGA-A and SGA-B/C) will be assessed by Kappa statistics and C-statistics respectively.

A multivariate logistic regression will be used to generate the adjusted odds ratios that quantify the association between high-mNUTRIC, malnutrition, and their combination (mNUTRIC ≥ 5 and SGA-B/C) with hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old who had ≥ 24 hours length of stay in the ICU
* received a nutrition assessment (SGA) from a dietitian within 48 hours of admission to the ICU

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU between August-2015 and October-2016 will be enrolled.
Sampling Method: Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | Up to one year after admission to the ICU
  All patients will be followed until discharge or death

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coltman A, Peterson S, Roehl K, Roosevelt H, Sowa D. Use of 3 tools to assess nutrition risk in the intensive care unit. JPEN J Parenter Enteral Nutr. 2015 Jan;39(1):28-33. doi: 10.1177/0148607114532135. Epub 2014 Apr 18. PMID 24748598